CLINICAL TRIAL: NCT01025622
Title: Phase 1 Study of Intrahepatic Reinfusion of Highly Purified CD133+ Stem Cells in Patients With End-Stage Liver Disease
Brief Title: Intrahepatic Reinfusion of CD133+ Stem Cells in Cirrhotic Patients
Acronym: Cirrhosis133
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Roberto M. Lemoli, MD, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-011783-10
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Liver Cirrhosis
Keywords: Stem Cells; Liver Cirrhosis; Cell Therapy
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: autologous highly purified CD133+ stem cells (SCs) — Intrahepatic reinfusion in cirrhotic patients

SUMMARY:
OBJECTIVE(S): Primary:

To assess the safety of the intrahepatic reinfusion of increasing numbers of autologous highly purified CD133+ stem cells (SCs) to patients with end-stage liver disease. Safety will be evaluated as the incidence of adverse event (graded according to WHO) and clinically significant abnormal laboratory value following reinfusion of SCs.

Secondary:

To assess the feasibility of the immunomagnetic selection of autologous CD133+ cells collected with leukapheresis from the peripheral blood (PB) of patients with end-stage liver disease, previously mobilized with G-CSF. To assess the effects of the intrahepatic reinfusion of highly purified CD133+ cells on residual hepatic function of the patients.

STUDY DESIGN:

Twelve patients will be enrolled. At first, G-CSF at 7.5µg/Kg/b.i.d. will be administered subcutaneously (sc) from day 1 until the completion of peripheral blood stem cells (PBSC) collection. Harvest of bone marrow (BM)-derived PBSC will begin on day + 4 only if the concentration of CD133+ cells is > 8/uL and will be continued until the collection of the target cell dose: 0.5 x 106 CD133+ cells/Kg for the first 2 cohorts of patients; 1 x 106 CD133+ cells/Kg for cohort 3 and 2 x 106 CD133+ cells/Kg for cohort 4 (see below for definitions). PB mononuclear cells obtained from mobilized standard-volume leukapheresis will be incubated with Macs colloidal superparamagnetic CD133 microbeads and CliniMacs device will be used for the positive selection of CD133+ cells under good manufacturing practice (GMP) conditions. Cryopreservation and storage in liquid nitrogen will be performed according to standard procedures. At least 4 weeks after SC mobilization and collection, up to 40 mL of single cell suspension of highly purified autologous CD133+ cells, obtained after rapid thawing, will be infused through the hepatic artery by transfemoral or transbrachial arteriography. Infusion time will be lower than 15ml/min to avoid thrombi formation. The entire procedure will be performed under anesthesiological control. According to modified Fibonacci's increment rule, highly purified G-CSF-mobilized CD133+ cells will be administered to patients starting from 5x104/Kg patient's body weight and increased every 3 patients. The maximum infused cell dose will be 1x106/kg. G-CSF at 5µg/Kg/day will be administered sc for 3 days after the reinfusion of SCs (day 0 to day +2).

DETAILED DESCRIPTION:
TITLE: Phase I study of intrahepatic reinfusion of highly purified CD133+ stem cells in patients with end-stage liver disease.

PRINCIPAL INVESTIGATOR: Roberto M. Lemoli, MD CO-INVESTIGATORS: Pietro Andreone, MD, Francesca Bonifazi, MD; Lucia Catani, BS; Antonia D'Errico, MD; Michelangelo Fiorentino, MD; Valeria Giudice, MD; Annagiulia Gramenzi, MD; Elisabetta Loggi, BS; Stefania Lorenzini, MD; Francesco Losinno, MD; Maria Rosa Motta, BS; Simonetta Rizzi, BS; Cristina Rossi, MD.

STUDY CENTER: Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi, Bologna - Italia, Unità Operativa di Ematologia in collaboration with:

Unità Operativa di Semeiotica Medica Unità Operativa di Anatomia e Istologia Patologica Unità Operativa di Immunoematologia e Trasfusionale Unità Operativa di Radiologia

CLINICAL PHASE: Phase I

OBJECTIVE(S): Primary:

To assess the safety of the intrahepatic reinfusion of increasing numbers of autologous highly purified CD133+ stem cells (SCs) to patients with end-stage liver disease. CD133+ SCs will be previously collected and cryopreserved after mobilization with granulocyte-colony stimulating factor (G-CSF) and leukapheresis. Safety will be evaluated as the incidence of adverse event (graded according to WHO) and clinically significant abnormal laboratory value following reinfusion of SCs.

Secondary:

To assess the feasibility of the immunomagnetic selection of autologous CD133+ cells collected with leukapheresis from the peripheral blood (PB) of patients with end-stage liver disease, previously mobilized with G-CSF.

To assess the effects of the intrahepatic reinfusion of highly purified CD133+ cells on residual hepatic function of the patients. In particular, the following values will be monitored: synthesis of proteins (albumin), synthesis of factors of the coagulation (prothrombin time, INR, fibrinogen, antithrombin III, thromboplastin time), bilirubinemia, proliferative activity, biosynthetic capacity (cholesterol, pseudocholinesterase).

To assess the effects of the treatment on the production of selected cytokines during the administration of G-CSF and after the intrahepatic reinfusion of highly purified CD133+ SCs to patients with end-stage liver disease.

STUDY DESIGN:

Twelve patients will be enrolled within 18-24 months in the dose-finding phase. The study has been designed as follows: at first, G-CSF (Lenograstim, Aventis Pharma or Filgrastim, Amgen) at 7.5µg/Kg/b.i.d. will be administered subcutaneously (sc) from day 1 until the completion of peripheral blood stem cells (PBSC) collection. Harvest of bone marrow (BM)-derived PBSC will begin on day + 4 only if the concentration of CD133+ cells is > 8/uL and will be continued until the collection of the target cell dose: 0.5 x 106 CD133+ cells/Kg for the first 2 cohorts of patients; 1 x 106 CD133+ cells/Kg for cohort 3 and 2 x 106 CD133+ cells/Kg for cohort 4 (see below for definitions). PB mononuclear cells obtained from mobilized standard-volume leukapheresis will be incubated with Macs colloidal superparamagnetic CD133 microbeads (Miltenyi Biotec, Bergisch Gladbach, Germany) and CliniMacs device will be used for the positive selection of CD133+ cells under good manufacturing practice (GMP) conditions (see attachments). Cryopreservation and storage in liquid nitrogen will be performed according to standard procedures (see attachments).

At least 4 weeks after SC mobilization and collection, up to 40 mL of single cell suspension of highly purified autologous CD133+ cells, obtained after rapid thawing, will be infused through the hepatic artery by transfemoral or transbrachial arteriography. Infusion time will be lower than 15ml/min to avoid thrombi formation. The entire procedure will be performed under anesthesiological control. The intrahepatic route of administration is deemed necessary to avoid the potential massive spleen trapping of CD133+ cells after conventional intravenous reinfusion in cirrhotic patients. Within 24 hours from the procedure, a doppler ultrasonography of the celiac trunk will be performed to exclude thrombotic events of the mesenteric district.

According to modified Fibonacci's increment rule, highly purified G-CSF-mobilized CD133+ cells will be administered to patients starting from 5x104/Kg patient's body weight and increased every 3 patients. The maximum infused cell dose will be 1x106/kg (see below). Lenograstim or Filgrastim at 5µg/Kg/day will be administered sc for 3 days after the reinfusion of SCs (day 0 to day +2) for their expansion and to induce a selective proliferative advantage of reinfused cells in vivo.

NUMBER OF PATIENTS AND TIME FRAME: Twelve patients will be enrolled within 18-24 months in the dose-finding phase.

DIAGNOSIS AND INCLUSION CRITERIA: Signed informed consent. Age >18. Karnofsky score > 70% or WHO <1. Adequate renal (serum creatinine < 2 mg/dl) and pulmonary (Sat O2 > 96%) function. Diagnosis of advanced, end-stage liver disease defined by a Mayo Model for End Stage Liver Disease (MELD) score between 17 and 25.

Patients with the following liver disease etiologies will be enrolled in the study: chronic viral hepatitis B, chronic viral hepatitis C, chronic viral hepatitis D, alcoholic cirrhosis, primary sclerosing cholangitis, primary biliary cirrhosis, Wilson's disease, genetic haemochromatosis or iron over-load cirrhosis, cirrhosis due to non alcoholic steato-hepatitis. Patients with alcoholic liver cirrhosis should have withdrawn alcohol active consumption to be enrolled in the study.

Eligibility for orthotopic liver transplantation (OLT) is not a contraindication to enter in the clinical study. Patients in waiting list for OLT transplantation will not be withdrawn and will be transplanted as soon as a suitable donor will become available. Their MELD score will remain that recorded prior SCs infusion in case of improvement following the experimental procedure.

The presence of cirrhosis related symptoms, like ascites, peripheral edema, recurrent gastrointestinal tract bleeding, recurrent encephalopathy do not represent major contraindications to be enrolled into the study. The patients may be considered eligible when clinically stable.

EXCLUSION CRITERIA: HIV positivity. Pregnant or nursing females. Current uncontrolled infection. Intercurrent organ damage. Diagnosis of hepatocarcinoma. Complete portal thrombosis. Severe impairment of coagulative function (PT< 30%, INR>2.5, Platelets < 40x109/L) that would contraindicate artheriography. Grade IV splenomegaly.

Budd-Chiari Syndrome with sovrahepatic vein thrombosis and cirrhosis of unknown origin will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >18 years
* Karnofsky score >70% or WHO <1
* Adequate renal (serum creatinine < 2 mg/dl) and pulmonary (Sat O2 >96%) function
* Diagnosis of advanced, end-stage liver disease defined by a Mayo Model for End Stage Liver Disease (MELD) score between 17 and 25. Patients with the following liver disease etiologies will be enrolled in the study: chronic viral hepatitis B, chronic viral hepatitis C, chronic viral hepatitis D, alcoholic cirrhosis (without alcohol active consumption), primary sclerosing cholangitis, primary biliary cirrhosis, Wilson's disease, genetic hemochromatosis or iron over-load cirrhosis, cirrhosis due to non alcoholic steato-hepatitis.

Eligibility for orthotopic liver transplantation (OLT) is not a contraindication to enter in the clinical study. Patients in waiting list for OLT transplantation will not be withdrawn and will be transplanted as soon as a suitable donor will become available.Their MELD score will remain that recorded prior SCs infusion in case of improvement following the experimental procedure.

The presence of cirrhosis related symptoms, like ascites, peripheral edema, recurrent gastrointestinal tract bleeding, recurrent encephalopathy do not represent major contraindications to be enrolled into the study.

The patients may be considered eligible when clinically stable.

Exclusion Criteria:

* HIV positivity
* Pregnant or nursing females
* Current uncontrolled infection
* Intercurrent organ damage
* Diagnosis of hepatocarcinoma
* Complete portal thrombosis
* Severe impairment of coagulative function (PT< 30%, INR>2.5, Platelets < 40x109/L) that would contraindicate arteriography
* Grade IV splenomegaly
* Budd-Chiari Syndrome with sovrahepatic vein thrombosis and cirrhosis of unknown origin will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events (graded according to WHO). Incidence of clinically significant abnormal laboratory values following reinfusion of highly purified CD133+ cells. | 1 year

SECONDARY OUTCOMES:
Effects of the intrahepatic reinfusion of highly purified CD133+ SCs on residual hepatic function of the patients: Child-Turcotte-Pugh and MELD score. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roberto M Lemoli, MD, Principal Investigator — University of Bologna
Locations (2):
- Italy (2):
  - Azienda Ospedaliera-Universitaria, Policlinico S. Orsola-Malpighi,, Bologna
  - Azienda Ospedaliera-Universitaria, Policlinico S. Orsola-Malpighi, Bologna

REFERENCES:
- See also: Local ethics committee — http://www.aosp.bo.it/content/comitato-etico